CLINICAL TRIAL: NCT05016206
Title: A Single Ascending Dose, Randomized, Double-Blind, Double-Dummy, Placebo- and Positive Controlled Study to Evaluate the Effect of ACH-0144471 on the QT Interval in Healthy Adult Subjects
Brief Title: A Study of the Cardiac Effects of Danicopan in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ACH471-013
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: Danicopan; ALXN2040; ACH-0144471; Electrocardiogram; QT Interval; Concentration-QT
MeSH Terms: interventions — danicopan; rhoA GTP-Binding Protein; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: This was a double-dummy, placebo- and positive-controlled study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (ABC) (Experimental): Treatment Sequence ABC - Participants received all 3 doses of danicopan in ascending fashion over 3 periods:
  Treatment A (Period 1): Danicopan 400 milligrams (mg) and moxifloxacin-matching placebo.
  Treatment B (Period 2): Danicopan 800 mg and moxifloxacin-matching placebo.
  Treatment C (Period 3): Danicopan 1200 mg and moxifloxacin-matching placebo.
  Interventions: Drug: Danicopan; Drug: Moxifloxacin-matching Placebo
- Control Arm (EFG and IJK) (Placebo Comparator): Participants received 1 of 2 treatment sequences (Treatment Sequence EFG or Treatment Sequence IJK) over 3 periods:
  Treatment E (Period 1): Danicopan-matching placebo (400 mg) and moxifloxacin-matching placebo.
  Treatment F (Period 2): Danicopan-matching placebo (800 mg) and moxifloxacin 400 mg.
  Treatment G (Period 3): Danicopan-matching placebo (1200 mg) and moxifloxacin-matching placebo.
  Treatment I (Period 1): Danicopan-matching placebo (400 mg) and moxifloxacin 400 mg.
  Treatment J (Period 2): Danicopan-matching placebo (800 mg) and moxifloxacin-matching placebo.
  Treatment K (Period 3): Danicopan-matching placebo (1200 mg) and moxifloxacin 400 mg.
  Interventions: Drug: Moxifloxacin-matching Placebo; Drug: Danicopan-matching placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Danicopan — Danicopan tablets administered as a single oral dose.
  Other Names: ALXN2040; ACH-0144471 (formerly); ACH-4471; ACH4471; 4471
  Arms: Treatment Arm (ABC)
Drug: Moxifloxacin-matching Placebo — Moxifloxacin-matching placebo was administered as a single oral dose.
Drug: Danicopan-matching placebo — Danicopan-matching placebo was administered as a single oral dose.
  Arms: Control Arm (EFG and IJK)
Drug: Moxifloxacin — Moxifloxacin 400 mg was administered as a single tablet oral dose.
  Other Names: Avelox
  Arms: Control Arm (EFG and IJK)

SUMMARY:
This was a randomized, double-blind, double-dummy, placebo- and positive-controlled, 2-arm (Treatment Arm and Control Arm), parallel study to evaluate the effect of ACH-0144471 (danicopan) on the QT interval in healthy adult participants.

DETAILED DESCRIPTION:
Participants randomized to the Treatment Arm received all 3 doses of danicopan in a single ascending fashion over 3 periods (Treatment Sequence ABC). A single oral dose of danicopan was administered with a moxifloxacin-matching placebo on Day 1 of each period.

Participants randomized to the Control Arm were further randomized to receive 1 of 2 treatment sequences (Treatment Sequences EFG or IJK). A single oral dose of danicopan-matching placebo was administered with moxifloxacin or with moxifloxacin-matching placebo, as per the assigned randomization scheme, on Day 1 of each period.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index in the range of 18.0 to 32.0 kilograms (kg)/meter squared, inclusive, with a minimum body weight of 50 kg at screening.
* Female participants must have been of nonchildbearing potential.
* Nonsterile male participants must have agreed to abstinence or used a highly effective method of contraception.
* No clinically significant history or presence of electrocardiogram findings at screening and check-in.

Key Exclusion Criteria:

* Evidence of any clinically significant deviation from normal in clinical laboratory evaluations.
* History of any medical or psychiatric condition or disease that might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
* History or presence of drug or alcohol abuse within 2 years prior to first dosing; current tobacco/nicotine user or a positive cotinine test at screening; positive for alcohol and/or drugs-of-abuse screen at screening or first check-in.
* Any previous procedure that could alter absorption or excretion of orally administered drugs.
* A history of significant multiple and/or severe allergies or had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs.
* Body temperature ≥ 38°Celsius on Day -2 or Day 1 prior to first dosing; history of febrile illness, or other evidence of infection, within 14 days prior to first dosing.
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives (if known) or 30 days before first dosing, whichever was longer.
* Donation of whole blood from 3 months before first dosing, or of plasma from 30 days before first dosing; received blood products within 6 months before first dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected Change From Baseline In QTc Intervals (ddQTc) For Danicopan | Pre-dose through 24 hours post-dose

SECONDARY OUTCOMES:
Change From Baseline In Heart Rate (HR) For Danicopan | Pre-dose through 24 hours post-dose
Change From Baseline In QT Interval For Danicopan | Pre-dose through 24 hours post-dose
Change From Baseline In Pulse Rate (PR) For Danicopan | Pre-dose through 24 hours post-dose
Change From Baseline In RR Interval For Danicopan | Pre-dose through 24 hours post-dose
Change From Baseline In QRS Interval For Danicopan | Pre-dose through 24 hours post-dose
ddQTcF Of Moxifloxacin | Pre-dose through 24 hours post-dose
Treatment-emergent T-wave Morphology Abnormalities And Pathologic U-waves | Pre-dose through 24 hours post-dose
Area Under The Plasma Concentration Versus Time Curve From Time 0 To 24 Hours Post-dose (AUC0-24) Of Danicopan | Pre-dose through 24 hours post-dose
Maximum Observed Plasma Concentration (Cmax) Of Danicopan | Pre-dose through 24 hours post-dose
Time To Reach The Maximum Observed Plasma Concentration (Tmax) Of Danicopan | Pre-dose through 24 hours post-dose
Number Of Participants Experiencing Treatment-emergent Adverse Events | Day 1 (postdose) through follow-up visit (14 [+/- 2] days after last study drug administration)]

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes